CLINICAL TRIAL: NCT02608892
Title: Caring for Babies During the Newborn Screening Blood Test: How do Parents Help? A Pilot RCT
Brief Title: Caring for Babies During the Newborn Screening Blood Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Denise Harrison, Chair in Nursing Care of Children, Youth and Families, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15/176X
Record Dates: First submitted 2015-11-11; First posted 2015-11-20 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Pain
Keywords: Breastfeeding; Skin to skin care; Sucrose; Newborn screening; Blood test; Neonate; Infant; Knowledge translation
MeSH Terms: conditions — Pain; Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): BSweet2Babies video
  Interventions: Behavioral: BSweet2Babies video
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: BSweet2Babies video — Mothers (and partners if possible) will view the brief BSweet2Babies video on electronic notebooks in French or English, as per parent/s' preference.
  Arms: Intervention

SUMMARY:
Newborn infants have blood work procedures in their first days of life that cause pain, distress and physiological changes. Breastfeeding (BF), skin to skin care (SSC), or giving sweet solutions (sucrose or glucose) has been shown to be effective for reducing babies' pain. However, recent studies of neonatal pain management practices demonstrate infrequent use of these strategies. There is a need for parent-targeted interventions, to support parents' involvement in comforting their infants during painful procedures. This pilot RCT will inform all aspects of a full-scale trial and will evaluate the effectiveness of the BSweet2Babies video when shown to parents of newborns prior to newborn screening, on subsequent use of effective pain reduction strategies during the newborn screening blood test. The participants will be randomized to either the control group (usual care), or to the intervention group and will be shown the brief BSweet2Babies video on caring for infants during blood work. The intervention group will be asked to complete a second survey after viewing the video. To evaluate the use of BF, SSC, or sucrose during newborn screening, the research assistant will collect data from the electronic medical record.

DETAILED DESCRIPTION:
Background: Newborn infants have blood work procedures for screening and medical monitoring in their first days of life that cause pain, distress and physiological changes. Breastfeeding (BF), skin to skin care (SSC), or giving small amounts of sweet solutions (sucrose or glucose) with or without a pacifier, effectively and safely reduce pain in newborn infants during painful procedures. However, recent studies of neonatal pain management practices demonstrate infrequent use of these strategies. There is a clear need for developing and testing acceptable parent-targeted interventions, alongside health care provider-targeted knowledge translation (KT) interventions, to support parents' involvement in comforting their infants during painful procedures. To address this knowledge to action (KTA) gap, Denise Harrison's Be Sweet to Babies team developed the BSweet2Babies video, which shows parents the effectiveness of BF, SSC, and sucrose during infant bloodwork and how they can use and advocate for these pain treatment strategies.

Objectives: To conduct a pilot randomized controlled trial (RCT) that will inform all aspects of a full-scale trial of the parent-targeted BSweet2Babies knowledge to action (KTA) intervention. The objective of the full scale trial will be to evaluate the effectiveness of the BSweet2Babies video when shown to parents of newborns prior to newborn screening, on subsequent use of effective pain reduction strategies during the newborn screening blood test.

Study design and methods: This study is a pilot 2-armed RCT that will enroll 100 parents in the mother baby unit at The Ottawa Hospital. Following consent, the research assistant will randomize parents to one of two groups: the intervention group (viewing the BSweet2Babies video prior to their baby's newborn screening blood test) or the control group (no intervention). Parents in both groups will complete a brief baseline survey to establish previous knowledge and use of pain management strategies. Participants in the intervention group will subsequently view the 5 minute BSweet2Babies video. Lastly, participants in the intervention group will be asked to complete a second online survey after viewing the video. To evaluate the use of BF, SSC or sucrose during newborn screening, the study research assistant will collect the data from the baby's electronic medical record.

Outcome Measures: The primary outcome is the use of BF, SSC or sucrose during newborn screening measured using data from the electronic medical records. The secondary outcomes are: i) feasibility of recruiting parents and showing the video prior to the infants' newborn screening; ii) effectiveness (i.e. did the video influence intent to use/advocate for one of the strategies); iii acceptability (i.e. would they recommend the video to other parents and suggested improvements to the video). The secondary outcomes will be measured with the online survey.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the mother baby unit;
* understands English or French, and
* their infant is eligible to receive breastfeeding, skin to skin care, or sucrose during newborn screening.

Exclusion Criteria:

- N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Harrison, RN, PhD, Principal Investigator — Children's Hospital of Eastern Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between May and August 2016, at a mother-baby unit in Ontario, Canada.
Pre-assignment Details: No enrolled participants were excluded from the study before assignment to groups.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 51 | 49
Completed | 50 | 49
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Viewed the BeSweet2Babies video.
- Control Group: Received usual care.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (5) | 32.9 (6) | 32.3 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 30 | 26 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Management Used During Newborn Screening Blood Test
Description: Use of any pain management: breastfeeding or skin to skin care or sucrose
Time Frame: Within 48 hours of viewing video intervention
Population: One participant was lost to follow-up in the intervention group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 50 | 49
Participants | 30 | 33
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority — Use of pain management during newborn screening was described using frequency and proportion and expressed as an absolute difference in proportions with 95% confidence interval; Absolute difference in proportions = -7.4, 95% CI 2-sided [-26.2 to 11.5]

2. Secondary Outcome: The Proportion of Parents Who Intend to Use or Advocate for at Least One of the Pain Management Strategies During Future Procedures
Description: Parents who viewed the intervention video will be asked one survey question about if they intend to use or advocate for breastfeeding, skin to skin care and/or sucrose during future procedures (yes/no)
Time Frame: Within 24 hours after viewing video intervention
Population: All 51 participants in the intervention group provided data for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: Only those in the intervention group (who viewed the BeSweet2Babies video) were asked.
Arm/Group | Intervention Group
Number analyzed (Participants) | 51
Participants
  Yes | 51
  No | 0

3. Secondary Outcome: Proportion of Parents Who Intend to Recommend the Video to Other Parents
Description: Parents who viewed the intervention video will be asked one survey question about if they intend to recommend the video to other parents (yes/no)
Time Frame: Within 24 hours after viewing video intervention
Population: All 51 participants in the intervention group provided data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 51
Participants
  Yes | 51
  No | 0

4. Secondary Outcome: Proportion of Parents Who Perceive the Duration of the Video as Acceptable
Description: Parents who viewed the intervention video will answer one survey question about their perception of whether the 5-minute video was of appropriate duration (too long/too short/just right)
Time Frame: Within 24 hours after viewing video intervention
Population: All 51 participants in the intervention group provided data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 51
Participants
  Just right | 49
  Too short | 0
  Too long | 2

ADVERSE EVENTS:
Time Frame: Up to time of patient discharge from unit (i.e. up to 24-48 hours)
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 0/51 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes